CLINICAL TRIAL: NCT04523142
Title: A Phase 3, Multi-center, Open-label, Single-arm Clinical Trial to Assess the Long-term Safety and Tolerability of Topical CyclASol® for the Treatment of Dry Eye Disease in Subjects Who Completed the Clinical Trial CYS-004
Brief Title: CyclASol for the Treatment of Signs and Symptoms of Dry Eye Disease in Subjects Who Completed CYS-004
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYS-005
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-08

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CyclASol Ophthalmic Solution (Experimental): Cyclosporine A solution in vehicle
  Interventions: Drug: CyclASol Ophthalmic Solution

INTERVENTIONS:
Drug: CyclASol Ophthalmic Solution — Cyclosporine A solution in vehicle

SUMMARY:
The objective of this trial is to evaluate safety and tolerability of CyclASol during long-term use in subjects with Dry Eye Disease.

DETAILED DESCRIPTION:
Phase 3 multicenter, open-label, single-arm clinical trial to evaluate the safety, tolerability and efficacy of CyclASol in subjects with signs and symptoms of Dry Eye Disease. Subjects who completed the trial CYS-004, had a subject-reported history of dry eye in both eyes and met all other study eligibility criteria were dosed CyclASol bilaterally BID for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the clinical trial CYS-004 and habe been compliant with trial procedures
* Signed ICF (Informed Consent Form)
* Subject-reported history of DED in both eyes
* Ability and willingness to follow instructions, including participation in all study assessments and visits

Exclusion Criteria:

* Early termination of CYS-004
* Clinically significant slit-lamp findings or ocular conditions that require prescriptive medical treatment and/or in the opinion of the investigator may interfere with trial parameters
* Have a history of herpetic keratitis;
* Have an ocular or periocular malignancy;
* Be unwilling to avoid wearing contact lenses during the trial;
* Have any planned ocular or eyelid surgeries during the trial period
* Be a woman who is pregnant, nursing or planning a pregnancy
* Unwillingness to submit a urine pregnancy test at all onsite visits if of childbearing potential
* Women of childbearing potential not using an acceptable means of contraception
* Presence of known allergy and/or sensitivity to the study drug or its components
* Be currently using an investigational drug or device or have used an investigational drug or device within 60 days before Visit 1 other than for CYS-004
* Have a condition or be in a situation (eg language barrier) which the investigator feels may put the subject at significant risk,may confound the trial results, or may interfere with the subject's participation in the trial significantly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Kroesser, PhD, Study Director — Novaliq GmbH
Locations (14):
- United States (14):
  - CYS-005 Investigational Site, Los Angeles, California
  - CYS-005 Investigational Site, Newport Beach, California
  - CYS-005 Investigational Site, Carmel, Indiana
  - CYS-005 Investigational Site, Louisville, Kentucky
  - CYS-005 Investigational Site, Andover, Massachusetts
  - CYS-005 Investigtional Site, Raynham, Massachusetts
  - CYS-005 Investigational Site, Henderson, Nevada
  - CYS-005 Investigational Site, Raleigh, North Carolina
  - CYS-005 Investigational Site, Shelby, North Carolina
  - CYS-005 Investigational Site, Fargo, North Dakota
  - CYS-005 Investigational Site, Cranberry Township, Pennsylvania
  - CYS-005 Investigational Site, Memphis, Tennessee
  - CYS-005 Investigational Site, Layton, Utah
  - CYS-005 Investigational Site, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wirta DL, Galor A, Aune CA, Vollmer PM, Liang E, Meides AS, Krosser S. Long-Term Safety and Efficacy of a Water-Free Cyclosporine 0.1% Ophthalmic Solution for Treatment of Dry Eye Disease: ESSENCE-2 OLE. Cornea. 2024 May 21;44(6):692-700. doi: 10.1097/ICO.0000000000003567. PMID 38771801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single arm, open label
Groups:
- CyclASol Ophthalmic Solution: Cyclosporine A solution in vehicle
  CyclASol Ophthalmic Solution: Cyclosporine A solution in vehicle (one drop per eye BID).
Period: Overall Study
Arm/Group | CyclASol Ophthalmic Solution
Started | 202 (202 participants were enrolled. Two participants were lost to follow-up directly after Visit 1. The safety population comprised 200 participants.)
Completed | 175
Not Completed | 27

BASELINE CHARACTERISTICS:
Population: 202 participants were enrolled. Two participants were lost to follow-up directly after Visit 1. The safety population comprised 200 participants.
Arm/Group | CyclASol Ophthalmic Solution
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 175
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 153
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any Adverse Events
Description: An adverse event was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not the event was considered drug related. 200 participants from the safety set were analyzed.
Time Frame: 12 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | CyclASol Ophthalmic Solution
Number analyzed (Participants) | 200
Participants | 97

ADVERSE EVENTS:
Time Frame: Data were collected over 52 weeks
Description: Ocular and non-ocular AEs were the primary safety endpoints in this study. An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not the event was considered drug related.
Arm/Group | CyclASol Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 4/200
Other Adverse Events (participants affected / at risk) | 13/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyclASol Ophthalmic Solution (N=200)
Transient ischemic attach (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CyclASol Ophthalmic Solution (N=200)
Instillation site pain (Eye disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04523142/Prot_SAP_000.pdf